CLINICAL TRIAL: NCT02117050
Title: RESOunD: REbif Satisfaction On Discontinuing Oral Dimethyl Fumarate. A 24-week, Prospective, Open-label, Multicenter Trial Evaluating Treatment Satisfaction in Subjects With Relapsing Forms of Multiple Sclerosis Following Treatment Change From Tecfidera™ to Rebif® 44 mcg Subcutaneously (sc) Three Times Weekly (Tiw)
Brief Title: RESOunD: REbif Satisfaction On Discontinuing Oral Dimethyl Fumarate
Acronym: RESOunD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment challenges
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR200136-586
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Rebif ®; Tecfidera ™; treatment change
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

ARMS (1):
- Rebif® via Rebidose® auto-injector (Experimental)
  Interventions: Drug: Rebif®

INTERVENTIONS:
Drug: Rebif® — Rebif® will be administered subcutaneously three times a week at a dose of 8.8 to 44 microgram (mcg) in initial titration schedule (5 weeks), followed by Rebif® 44 mcg subcutaneously three times a week by using Rebif® Rebidose® auto-injector device till Week 24.
  Other Names: interferon-beta-1a

SUMMARY:
This is a Phase IV, prospective, open-label, multi-center trial to assess the treatment satisfaction in patients with relapsing forms of Multiple Sclerosis (MS) who are currently being treated with, but are considering discontinuing treatment with Tecfidera™.

ELIGIBILITY:
Key inclusion Criteria:

* Diagnosis of relapsing form of MS
* Have declared a desire/plan to discontinue treatment with Tecfidera due to tolerability issues and/or lack of efficacy
* Expanded Disability Status Scale (EDSS) score 0 to 5.0 inclusive
* Other protocol defined inclusion criteria could apply

Key exclusion Criteria:

* Pregnant or lactating
* Significant renal or hepatic impairment or other significant disease that would compromise adherence and completion of the trial
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, MD, Study Director — EMD Serono, Inc., an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Call EMD Serono Medical Information for information on recruiting sites, Boston, Massachusetts, United States

REFERENCES:
- See also: The North American Research Committee on Multiple Sclerosis - Information about the PDDS Questionaire — http://www.narcoms.org/pdds

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was prematurely terminated due to enrollment issues. Only 1 subject was enrolled in this study, but did not receive any dose.
Groups:
- Rebif® Via Rebidose® Auto-injector: Rebif® was to be administered subcutaneously three times a week at a dose of 8.8 to 44 microgram (mcg) in initial titration schedule (5 weeks), followed by Rebif® 44 mcg subcutaneously three times a week by using Rebif® Rebidose® auto-injector device till Week 24.
Period: Overall Study
Arm/Group | Rebif® Via Rebidose® Auto-injector
Started | 1
Completed | 0
Not Completed | 1
Not completed — Subject Enrolled but not Dosed | 1

BASELINE CHARACTERISTICS:
Groups:
- Rebif® Via Rebidose® Auto-injector: Rebif® was to be administered subcutaneously three times a week at a dose of 8.8 to 44 mcg in initial titration schedule (5 weeks), followed by Rebif® 44 mcg subcutaneously three times a week by using Rebif® Rebidose® auto-injector device till Week 24.
Arm/Group | Rebif® Via Rebidose® Auto-injector
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex/Gender, Customized [Number; unit: subject]
  Prefers not to identify | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Treatment Satisfaction Score Determined by the Global Satisfaction Sub-scale of the Treatment Satisfaction Questionnaire for Medication (TSQM [Version II]) at Week 24
Description: The TSQM (Version II) is a validated tool that measures patient satisfaction with medical treatments using a 100-point scale. Global satisfaction sub-scale of TSQM was to be used to measure overall satisfaction with medication using a 100-point scale. Subject were to respond about their satisfaction or dissatisfaction with medication they are taking on a scale ranging from 0 to 100, where higher scores indicated greater satisfaction.
Time Frame: Baseline, Week 24
Population: The study enrolled only 1 subject who did not receive any dose. Thus, the data for primary endpoint was not collected.
Arm/Group | Rebif® Via Rebidose® Auto-injector
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline in Patient-Determined Disease Steps Questionnaire (PDDS) Score at Week 24
Description: PDDS questionnaire was to be used to assess the walking ability of subjects. Subjects were to describe their walking ability on scale ranging from 0 to 8, where 0 indicated normal walking and 8 indicated subject's condition as bedridden. Lesser score indicated better walking ability.
Time Frame: Baseline, Week 24
Population: The study enrolled only 1 subject who did not receive any dose. Thus, the data for secondary endpoint was not collected.
Arm/Group | Rebif® Via Rebidose® Auto-injector
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in Multiple Sclerosis Quality of Life-54 (MSQoL-54) Score at Week 24
Description: The MSQOL-54 is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument. MSQoL-54 is a 54 item questionnaire which covers 12 sub-scales along with two summary scores, and two additional single-item measures. The 12 sub-scales are: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, and sexual function. The 2 summary scores are the physical health composite summary and the mental health composite summary. The 2 additional single item measures are satisfaction with sexual function and change in health. Each of the 12 sub-scale scores, the 2 summary scores and 2 single item measures were to be converted into an overall Total Score ranging from 0-100, where higher scores indicated better health status.
Time Frame: Baseline, Week 24
Population: The study enrolled only 1 subject who did not receive any dose. Thus, the data for secondary endpoint was not collected.
Arm/Group | Rebif® Via Rebidose® Auto-injector
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in TSQM (Version II) - Total Score at Week 12 and Week 24
Description: The TSQM (Version II) is an 11-item validated tool that measures patient satisfaction with medical treatments using a 100-point scale. Total TSQM score was the average of individual sub-scale scores (effectiveness, side effects, convenience and global satisfaction) and ranged from 0 to 100, where higher scores indicated greater satisfaction.
Time Frame: Baseline, Week 12 and Week 24
Population: The study enrolled only 1 subject who did not receive any dose. Thus, the data for secondary endpoint was not collected.
Arm/Group | Rebif® Via Rebidose® Auto-injector
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in TSQM (Version II) - Medication Effectiveness, Side Effects, and Convenience Subscale Scores at Week 24
Description: The TSQM (Version II) is a validated tool that measures patient satisfaction with medical treatments using a 100-point scale. Effectiveness, side effects and convenience sub-scales of TSQM were to be used to measure overall satisfaction with medication. Subject were to respond about their satisfaction or dissatisfaction with medication they are taking in terms of effectiveness, side effects and convenience, each sub-scale ranging on a scale of 0 to 100, where higher scores indicated greater satisfaction.
Time Frame: Baseline, Week 24
Population: The study enrolled only 1 subject who did not receive any dose. Thus, the data for secondary endpoint was not collected.
Arm/Group | Rebif® Via Rebidose® Auto-injector
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in TSQM (Version II) - Global Satisfaction, Medication Effectiveness, Side Effects, and Convenience Subscale Scores at Week 12
Description: The TSQM (Version II) is a validated tool that measures patient satisfaction with medical treatments using a 100-point scale. Effectiveness, side effects, convenience and global satisfaction sub-scales of TSQM were to be used to measure overall satisfaction with medication. Subject were to respond about their satisfaction or dissatisfaction with medication they are taking in terms of effectiveness, side effects, convenience and global satisfaction, each sub-scale ranging on a scale of 0 to 100, where higher scores indicated greater satisfaction.
Time Frame: Baseline, Week 12
Population: The study enrolled only 1 subject who did not receive any dose. Thus, the data for secondary endpoint was not collected.
Arm/Group | Rebif® Via Rebidose® Auto-injector
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment- General Health (WPAI-GH) Questionnaire Score at Week 24
Description: WPAI-GH questionnaire is a subject reported quantitative assessment of general health conditions on productivity. The Total WPAI-GH score assessment was to be done on an 11-point scale ranging 0 to 10, with 0 indicating that health problems had no effect on work and 10 indicating that health problems completely prevented from working.
Time Frame: Baseline, Week 24
Population: The study enrolled only 1 subject who did not receive any dose. Thus, the data for secondary endpoint was not collected.
Arm/Group | Rebif® Via Rebidose® Auto-injector
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Number of Combined Unique Active (CUA) Lesions, New Time or Enlarging Constant 2 (T2) Lesions, and New Gadolinium Enhanced (Gd+) Time Constant 1 (T1) Lesions at Week 24
Time Frame: Baseline, Week 24
Population: The study enrolled only 1 subject who did not receive any dose. Thus, the data for secondary endpoint was not collected.
Arm/Group | Rebif® Via Rebidose® Auto-injector
Number analyzed (Participants) | 0

9. Secondary Outcome: Annualized Relapse Rate (ARR)
Description: A relapse is defined as new or recurrent neurologic symptoms not associated with fever or infection, lasting for at least 24 hours, and accompanied by new objective neurologic findings. Episodes indicated by neurologist as "relapse" in the subjects chart were to be recorded.
Time Frame: Week 24
Population: The study enrolled only 1 subject who did not receive any dose. Thus, the data for secondary endpoint was not collected.
Arm/Group | Rebif® Via Rebidose® Auto-injector
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The study was prematurely terminated due to one subject enrolled but not dosed. Thus, data for adverse events was not collected.
Arm/Group | Rebif® Via Rebidose® Auto-injector
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to enrollment issues. Only 1 subject was enrolled in this study, but did not receive any dose. Neither efficacy nor safety analysis was done for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study as a whole will be published prior to any individual investigator publications. It is required that copies of all papers, abstracts, articles, etc. that contain study data are to be forward to the Sponsor for review 30 days prior to submission for publication.